CLINICAL TRIAL: NCT04265729
Title: An Open-label, Explorative, Post Launch Study of Neocate Amino Acid-based Feeds to Evaluate Nutritional Status and Gastrointestinal Tolerance in Infants and Children With Complex Conditions
Brief Title: Neocate In Infants and Children With Complex Conditions
Acronym: NICC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MPR18TA23134
Record Dates: First submitted 2020-01-28; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Complex Conditions, Including Impairment of the GI Tract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single test product arm (Other): use of Neocate Infant and Junior marketed products (product type depending on subject's age and condition)
  Interventions: Dietary Supplement: Neocate Infant and Junior marketed products

INTERVENTIONS:
Dietary Supplement: Neocate Infant and Junior marketed products — use of Neocate Infant and Junior marketed products

SUMMARY:
Infants and young children up to 10 years of age with a complex condition involving the gastrointestinal tract are at risk of poor nutritional status, including faltering growth. Due to the complex condition, standard nutrition is often not tolerated and causes gastrointestinal symptoms.

Formulas in which protein is replaced by its smallest elements, amino acids are easier for the body to digest and absorb. These formulas might be tolerated better and reduce gastrointestinal symptoms in infants and young children with complex conditions.

The objectives of the present, exploratory study are to gain clinical evidence related to the nutritional status and gastrointestinal tolerance in infants and young children with complex conditions receiving Neocate as their primary source of nutrition. Additional objectives are to describe the nutritional and pharmacological management of these infants and young children. Study duration for each participant will be 52 weeks at maximum.

ELIGIBILITY:
Inclusion Criteria:

* Infants and young children aged from 0 up to and including 10 years of age.
* Severe impairment of at least 1 organ system
* Impairment of the gastrointestinal tract, i.e. gastrointestinal disease, congenital abnormality, surgical resection, or gastrointestinal dysfunction (including symptoms of gastrointestinal dysmotility or malabsorption).
* Receiving at least 75% of their energy intake from Neocate (Neocate Infant or Junior powdered (marketed) product) at the time of study entry (V1).
* Expected to receive at least 75% of their energy intake from the study product for at least 4 weeks from study entry (V1).
* Written informed consent provided by parents/guardians and assent by the child, if applicable, according to local law.

Exclusion Criteria:

* Infants born with a gestational age <37 weeks that are <40 weeks corrected age at the time of study entry (V1).
* Infants or children with endoscopically confirmed eosinophilic oesophagitis and prescribed an amino acid-based formula only for the management of the eosinophilic oesophagitis.
* Infants or children with a medical diagnosis that includes only (suspected) cow's milk allergy and/or multiple food allergy.
* Infants or children with renal dysfunction, e.g. acute or chronic kidney failure or kidney cancer.
* Infants or children with thyroid disorder or parathyroid disorder.
* Expected to receive parenteral nutrition during intervention from study entry (V1).
* Participation in any other studies involving investigational or marketed products concomitantly or within 1 month prior to study entry (V1).
* Investigator's uncertainty about the willingness or ability of the parents/guardians to comply with the protocol requirements.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Exploratory: Weight | 0 weeks
  Weight [in g/kg]
Exploratory: Weight | 4 weeks
  Weight [in g/kg]
Exploratory: Weight | 16 weeks
  Weight [in g/kg]
Exploratory: Weight | 52 weeks
  Weight [in g/kg]
Exploratory: Length | 0 weeks
  Length/height [in cm]
Exploratory: Length | 4 weeks
  Length/height [in cm]
Exploratory: Length | 16 weeks
  Length/height [in cm]
Exploratory: Length | 52 weeks
  Length/height [in cm]
Exploratory: head circumference | 0 weeks
  head circumference (for children <2 years of age) [in cm]
Exploratory: head circumference | 4 weeks
  head circumference (for children <2 years of age) [in cm]
Exploratory: head circumference | 16 weeks
  head circumference (for children <2 years of age) [in cm]
Exploratory: head circumference | 52 weeks
  head circumference (for children <2 years of age) [in cm]
Exploratory: Biochemical markers of nutritional status | 0 weeks
  Macronutrient, micronutrient and mineral levels in blood [in a.o. mmol/L]
Exploratory: Biochemical markers of nutritional status | 4 weeks
  Macronutrient, micronutrient and mineral levels in blood [in a.o. mmol/L]
Exploratory: Biochemical markers of nutritional status | 16 weeks
  Macronutrient, micronutrient and mineral levels in blood [in a.o. mmol/L]
Exploratory: Biochemical markers of nutritional status | 52 weeks
  Macronutrient, micronutrient and mineral levels in blood [in a.o. mmol/L]
Exploratory: Gastrointestinal tolerance | 0 weeks
  GastrointestinaI symptoms [none/mild/moderate/severe]
Exploratory: Gastrointestinal tolerance | 4 weeks
  GastrointestinaI symptoms [none/mild/moderate/severe]
Exploratory: Gastrointestinal tolerance | 16 weeks
  GastrointestinaI symptoms [none/mild/moderate/severe]
Exploratory: Gastrointestinal tolerance | 52 weeks
  GastrointestinaI symptoms [none/mild/moderate/severe]
Exploratory: Stool frequency | 0 weeks
  number of stools per day
Exploratory: Stool frequency | 4 weeks
  number of stools per day
Exploratory: Stool frequency | 16 weeks
  number of stools per day
Exploratory: Stool frequency | 52 weeks
  number of stools per day
Exploratory: Stool consistency | 0 weeks
  parent reported stool consistency using stool scales (scale depending on diaper use or not) with categories within the range hard to watery
Exploratory: Stool consistency | 4 weeks
  parent reported stool consistency using stool scales (scale depending on diaper use or not) with categories within the range hard to watery
Exploratory: Stool consistency | 16 weeks
  parent reported stool consistency using stool scales (scale depending on diaper use or not) with categories within the range hard to watery
Exploratory: Stool consistency | 52 weeks
  parent reported stool consistency using stool scales (scale depending on diaper use or not) with categories within the range hard to watery
Exploratory: Nutrient intake | 0 weeks
  calculated energy, protein and micronutrient levels from parent diary [in a.o. mg/d]
Exploratory: Nutrient intake | 4 weeks
  calculated energy, protein and micronutrient levels from parent diary [in a.o. mg/d]
Exploratory: Nutrient intake | 16 weeks
  calculated energy, protein and micronutrient levels from parent diary [in a.o. mg/d]
Exploratory: Nutrient intake | 52 weeks
  calculated energy, protein and micronutrient levels from parent diary [in a.o. mg/d]

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - GI Care for Kids, Atlanta, Georgia
  - Prisma Health - Upstate, Greenville, South Carolina
- Dr. von Haunersches LKinderspital, Munich, Germany
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No